CLINICAL TRIAL: NCT04217798
Title: A Single Arm, Prospective, Multicenter, Phase II Study to Evaluate the Efficacy and Safety of Niraparib Combined With Oral Etoposide in Platinum Resistant/ Refractory Recurrent Ovarian Cancer
Brief Title: Efficacy and Safety of Niraparib Combined With Oral Etoposide in Platinum Resistant/Refractory Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH1902001
Record Dates: First submitted 2019-12-09; First posted 2020-01-03 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2020-12

CONDITIONS: Ovarian Cancer
Keywords: platinum resistent/refractory, ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niparib combined with oral etoposide (Experimental): Subjects will received niraparib 200mg or 100mg alternate once daily and oral etoposide 50mg on day 1-20 of a 30-day cycle. Oral etoposide was administered for a maximum of 6-8 cycles. Treatment was continued until disease progression, patient withdrawal or unacceptable toxic effects.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Subjects will receive niraparib combined with oral etoposide (on day 1-20, every 30 days). After 6-8 cycles, oral etoposide will be terminated. Niraparib will be still given to subjects until disease progression, intolerable toxicity or withdrawal of informed consent.
  Other Names: oral etoposide

SUMMARY:
To evaluate the efficacy and safety of niraparib combined with oral etoposide in platinum resistant or platinum refractory recurrent ovarian cancer.

DETAILED DESCRIPTION:
This is a single arm, prospective, multicenter, phase II study to evaluate the efficacy and safety of PARP inhibitor niraparib combined with oral etoposide chemotherapy in women with platinum resistant or refractory recurrent ovarian cancer. Subjects will receive niraparib and oral etoposide in 30-day treatment cycles. After 6-8 cycles, oral etoposide will be discontinued. Subjects will receive niraparib alone until disease progression, intolerable toxicity or withdrawal of informed consent. The primary endpoint is progression free survival evaluated by Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Secondary endpoints include overall response rate , duration of response, disease control rate, CA125 response rate and safety.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before undertaking any study procedure.
* Female, age 18-70.
* Histologically confirmed FIGO stage III or IV non-mucinous epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
* No limitation of the BRCA mutation and HRD status.
* Platinum resistant or refractory recurrent disease.
* Subjects must have received at least 1 prior line of platinum-based chemotherapy regimen and no more than twice.
* Subjects must have measurable lesions with imaging evidence of disease progression (according to RECIST1.1 criteria); or without measurable/evaluable lesion (RECIST 1.1 criteria), but two consecutive cases of elevated CA125 > 2 times the upper limit of normal (> 70 U/ml) were detected.
* Life expectancy of more than 6 months.
* ECOG 0-1.
* Good organ function, including:

  * Bone marrow function: neutrophil count ≥1,500/µL, platelets ≥100,000/µL, hemoglobin ≥10 g/dL;
  * Hepatic function: total bilirubin ≤ 1.5 x upper limit of normal (ULN) or direct bilirubin ≤1.0 x ULN, AST and ALT ≤2.5 x ULN unless liver metastases are present, in which case they must be ≤5 x ULN;
  * Renal function: serum creatinine ≤1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥60 mL/min using the Cockcroft-Gault equation.
* Has a negative serum pregnancy test within 3 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 3 months after the last dose of study treatment, or is of non-childbearing potential. Non-childbearing potential is defined as follows (by other than medical reasons):

  * ≥45 years and <60 years of age and has not had menses for >1 year
  * ≥60 years of age
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation.
* Is able to adhere to the protocol.
* Has recovered from previous chemotherapy induced toxic side effects to ≤ grade 1 CTCAE or basal level, apart from ≤ grade 2 CTCAE peripheral neuropathy or hair loss symptoms at steady state.

Exclusion Criteria:

* Has a known hypersensitivity to the active or inactive ingredients of niraparib or compound which has similar chemical structure to niraparib.
* Has a known hypersensitivity to the active or inactive ingredients of etoposide or compound which has similar chemical structure to etoposide.
* prior PARP inhibitor therapy.
* Has symptomatic uncontrolled brain or leptomeningeal metastasis.
* Major surgery or chemotherapy within 3 weeks of starting the study or patient has not recovered from any effects of the surgery.
* Receive palliative radiotherapy encompassing > 20% of the bone marrow within 1 week of entering the study.
* Be diagnosed any invasive cancer other than ovarian cancer (apart from cured basal cell carcinoma and squamous cell carcinoma) within 2 years prior to study enrolment.
* Previously or currently diagnosed of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* Has other serious or uncontrolled disease.
* Has any disease, treatment and laboratory abnormality that may interfere the study results and affect the fully attendance of study. Or the subject is considered to be not suitable for the study by the investigator. Cannot receive platelet or red blood cell transfusion within 4 weeks of study drug administration.
* Pregnant, breastfeeding or expecting to conceive children during the study treatment period.
* Adjusted for QT interval (QTc) >470 msec.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Through study completion, an average of 1 year
  PFS is defined as the time from randomization to first disease progression by investigator assessment using RECIST 1.1 or death, from any cause, whichever comes first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Through study completion, an average of 1 year
  ORR is defined as the proportion of subjects who have a partial response (PR) or complete response (CR) to therapy according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Duration of Response (DOR) | Through study completion, an average of 1 year
  DOR is defined as the time from the first date of response until the date of first documented progression.
Disease Control Rate (DCR) | Through study completion, an average of 1 year
  DCR is defined as the proportion of subjects who have a complete response (CR), partial response (PR) and stable disease (SD) to therapy according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
CA125 Response Rate | Through study completion, an average of 1 year
  The proportion of subjects with a minimum 50% reduction in CA-125 serum levels lasting for ≥28 days relative to baseline CA-125 serum levels.
The frequency and severity of adverse events | Through study completion, an average of 1 year
  The frequency and severity of adverse events evaluated according to NCI CTCAE version 5.0 during subjects receiving the study treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing
  - Shandong Cancer Hospital, Jinan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou H, Liu Q, Zhang D, Li Q, Cao D, Cheng N, Wan X, Zhang Y, Feng F, Xiang Y, Yang J. Efficacy and safety of an oral combination therapy of niraparib and etoposide in platinum resistant/refractory ovarian cancer: a single arm, prospective, phase II study. Int J Gynecol Cancer. 2024 Nov 4;34(11):1761-1767. doi: 10.1136/ijgc-2024-005386. PMID 39074931